CLINICAL TRIAL: NCT05463445
Title: Multicenter Study of Clinical Characteristics and Management of Primary Sclerosing Cholangitis and IgG4-related Sclerosing Cholangitis in China.
Brief Title: Multicenter Observational Study of PSC and IgG4-SC in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, ma xiong, Principal Investigator, RenJi Hospital
Other Study IDs: SC2022CH001
Record Dates: First submitted 2022-07-14; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Primary Sclerosing Cholangitis; IgG4-related Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: patients diagnosed with Primary Sclerosing Cholangitis which met the PSC criteria according to The European Association for the Study of the Liver Clinical Practice Guidelines "Management of cholestatic liver diseases" in 2009.
  Interventions: Other: Only observation
- B: patients diagnosed with IgG4-related Sclerosing Cholangitis which met initially using the Japan Pancreas Society criteria and confirmed using HISORt criteria.
  Interventions: Other: Only observation

INTERVENTIONS:
Other: Only observation — No intervention is needed.

SUMMARY:
The investigators aimed to collect demographic features and clinical outcomes in patients diagnosed with PSC and IgG4-SC by utilizing participants database from multiple medical centers across Mainland China. Cross-sectional studies will focus on characterizing clinical presentations and validating diagnostic and prognostic models on Chinese PSC and IgG4-SC patients.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years old,
* Male or Female,
* Patients admitted in our medical centers which met the PSC criteria according to The European Association for the Study of the Liver Clinical Practice Guidelines "Management of cholestatic liver diseases" in 2009; or patients diagnosed with IgG4-SC which met initially using the Japan Pancreas Society criteria and confirmed using HISORt criteria.

Exclusion Criteria:

* Female subjects who is pregnant, breastfeeding or is considering being pregnant during the study;
* History of other malignancies, including hematological tumors, solid tumors except hepatobiliary system;
* History of infectious diseases, including hepatis A, B, C, E and tuberculosis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This program will be conducted in multiple medical centers among the major cities across Mainland China. The sample size of subjects will be 1000, including 500 patients with PSC and 500 patients with IgG4-SC.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of new occurrence of decompensated liver related events, malignancies, liver transplantation and liver-related death caused by PSC and IgG4-SC | 1 year
  describe the characteristics and clinical outcomes of PSC and IgG4-SC patients among multiple medical centers in China

CONTACTS AND LOCATIONS:
Locations (1):
- RenJi Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
After this observational study is recruited, we are welcome to share the basic demographics and clinical outcomes of recruited IPD.